CLINICAL TRIAL: NCT02557919
Title: Evaluation of the Smoking Cessation and Tobacco Use Exposure Patterns of Head Start Parents in Boston
Brief Title: Families Reduce Exposure to Smoke at Home
Acronym: FRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Truth Initiative (Other)
Responsible Party: Principal Investigator, Alan Geller, Senior Lecturer, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-0683
Record Dates: First submitted 2015-09-14; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Tobacco Use Cessation; Second Hand Tobacco Smoke
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing Training (Experimental): Staff at the intervention sites were trained in basic tobacco control and motivational interviewing. Two booster trainings were held over 6 months.
  Interventions: Other: Motivational Interviewing Training
- Usual Best Practice (Other): Staff at the usual best practice sites received basic tobacco control training.
  Interventions: Other: Usual Best Practice

INTERVENTIONS:
Other: Motivational Interviewing Training — 1.5 day training on Motivational Interviewing (MI) techniques plus 2 booster sessions to address real experiences using MI with families.
  Arms: Motivational Interviewing Training
Other: Usual Best Practice — .5 day training on tobacco control and emerging products.
  Arms: Usual Best Practice

SUMMARY:
This project proposes to evaluate the effectiveness of training Head Start staff to discuss tobacco use, shs reduction and cessation in their existing encounters with parents in reducing tobacco use and exposure. Understanding the facilitators and barriers to integrating the intervention into the Head Start system will support future efforts to address tobacco use and exposure in families with small children.

DETAILED DESCRIPTION:
Parental smoking increases children's risk of asthma, infectious illness, sudden infant death syndrome (SIDS), and other conditions. Accumulating evidence regarding the adverse effects of total smoke exposure (TSE) led the US Surgeon General to conclude that there is no safe level of TSE. Parents who smoke endanger themselves, put their children and spouses at risk for adverse health outcomes, and increase the chance of their children becoming smokers. However, many parents who smoke are undertreated for their tobacco addiction. Many parents who smoke are of the age where they have few contacts with primary care physicians and are often unexposed to counseling and pharmacotherapy offered to older patients. Strategically identifying sites where trained para-professionals routinely interact with parents who smoke is vital to making inroads in this high-risk population.

Involuntary secondhand smoke exposure (SHSe) in domestic environments is an entirely preventable public health threat that disproportionately burdens young children in communities of low socioeconomic position. Research has indicated that interventions to reduce SHSe for children delivered through child care settings have been effective. In addition, client-centered approaches, such as motivational interviewing, have been effective in helping parents to reduce levels of SHS in the home environment. Following guidelines from established agencies and organizations, we will also evaluate changes in smoking cessation rates among parents and staff comparing use prior to and after the training programs and subsequent family service worker to parent encounters.

Aim 1: Building on Action for Boston Community Development's (ABCD) current system efforts, support the development and implementation of system changes to accurately and efficiently document parental smoking and household tobacco use and exposure, using: i) intake form, ii) Individual Family Plan, and iii) electronic data system.

Aim 2: Collaborate with Legacy and University of Massachusetts (UMass) to train Head Start staff in skills for encouraging smoking cessation and on a smoke-free home intervention, to increase staff knowledge of second-hand smoke (SHS) effects and provide skills in Motivational Interviewing. This will enhance staff confidence in engaging with parents to assist in efforts to make a sustained quit attempt, reduce children's SHS exposure, and will provide structure to help staff determine how best to support families on issues of tobacco use, including referral to cessation services.

Aim 3: Evaluate the effectiveness of sites receiving the a) Motivational Interviewing intervention for family service workers, b) supervisor education, and c) boosters in decreasing parent smoking, reducing household tobacco use and children's SHS exposure, compared with sites receiving only basic tobacco information.

Aim 4: Evaluate the effectiveness of the smoking cessation intervention on the staff most intimately involved in parent counseling-namely, the family service workers who will attend the training program (s). We will evaluate their knowledge, attitudes, beliefs, and smoking practices as well as their confidence and skills in tobacco-related counseling.

ELIGIBILITY:
Inclusion Criteria:

* Parent Inclusion

  1. Parent of a child enrolled in an ABCD Early Head Start/Head Start Program
  2. Current smoker (1 or more cigarettes per day) and/or smoking is happening in or around (attached porches, patios, hallways) the family home by family members or regular visitors
  3. Able to complete a self-administered survey or request assistance from research staff
  4. Able to communicate in English or Spanish

Staff Inclusion

1. Staff member at one of the participating ABCD Head Start sites
2. Willing to consent to complete the staff survey

Exclusion Criteria:

* Parent Exclusion

  1. Unable or unwilling to consent to participate in this research
  2. No smoking is happening in or around the home

Staff Exclusion

1. Unwilling or unable to consent to complete the staff survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Tobacco quit attempts in the past 6 months (staff and parents) | Past 6 months
  Parents and staff will be surveyed to determine the number of quit attempts in the past 6 months.

SECONDARY OUTCOMES:
Home smoking ban implemented in the past 6 months | Past 6 months
  Parents will be surveyed to determine the number of home smoking bans implemented in the past 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Alan C Geller, RN, MPH, Principal Investigator — Harvard School of Public Health (HSPH)